CLINICAL TRIAL: NCT04236466
Title: Transverse Dento-skeletal Effects of Two Rapid Palatal Expansion Appliances in Cleft Lip and Palate Patients : A Randomized Clinical Trial
Brief Title: Transverse Dento-skeletal Effects of Two Rapid Palatal Expansion Appliances in Cleft Lip and Palate Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yomna Elfiky, teaching assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3-3-4
Record Dates: First submitted 2020-01-15; First posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Cleft Lip and Palate
Keywords: maxillary expansion
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hyrax group (Experimental): cleft lip and palate patients with hyrax appliance
  Interventions: Device: hyrax appliance
- haas group (Experimental): cleft lip and palate patients with haas appliance
  Interventions: Device: haas appliance

INTERVENTIONS:
Device: hyrax appliance — Hyrax will be constructed with bands on maxillary first molars and wire extending on palatal surfaces of teeth till the upper canines.
  Arms: hyrax group
Device: haas appliance — Haas will be constructed with bands on maxillary first molars and wire extending on palatal surfaces of teeth till the upper canines. Acrylic part will be added on palate
  Arms: haas group

SUMMARY:
Aim of the study: to compare the effect of Hyrax appliance and the Haas appliance improving the transverse skeletal and dental dimensions in cleft lip and palate patients during mixed dentition.

DETAILED DESCRIPTION:
•Steps in short Full records pre-treatment. Bands selection for upper first molars then construction of expansion appliances(Haas or Hyrax) . Delivery of appliances and instructions to the patients and their parents about their activation regimen 2 quarter turns in the morning and 2 in the evening.The posterior crossbite will be measured as the distance from the palatal cusp tips of upper first molars to central fossae of lower first molars then the needed time for expansion will be calculated .When the time calculated for correction ends, we will stop activation, we will take impressions for digital models to see if real expansion occurred or not and so testing the efficiency of the two appliances.

Afterthat, if correction was not yet achieved, activation of the appliances will continue till overcorrection at the molar region with the palatal cusp tip of the maxillary posterior teeth contacting the buccal cusp tip of the mandibular posterior teeth. We will then leave the appliance insitu for retention.

After 6 months from the first CBCT we will take a second CBCT to see any bony changes .

ELIGIBILITY:
Inclusion Criteria:

* (1) Mixed dentition; (2) Both males and females; (3) Lip repair performed between 3 and 6 months of age and palate repair performed between 12 and 24 months of age; (4) Presence of maxillary constriction and posterior crossbite and need for maxillary expansion previous to the secondary bone graft; (5) Permanent first maxillary molars present; (6) Good periodontal health; (7) No previous orthodontic treatment;

Exclusion Criteria:

* (1) Presence of a syndrome in companion with the present cleft defect (2) Previous secondary alveolar bone grafting (3)Taking medications affecting growth

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Tranverse dental changes | 3 months
  assessed on digital models by linear measurements (mm)
Tranverse dental changes | 6 months
  assessed on digital models by linear measurements(mm)
Tranverse skeletal changes | 6 months
  assessed on CBCT by linear and angular measurements(mm and angles)

SECONDARY OUTCOMES:
Maxillary and mandibular anteroposterior measurements | 3 months
  They will be measured on digital casts by linear measurements(mm)
Maxillary and mandibular anteroposterior measurements | 6 months
  They will be measured on digital casts by linear measurements(mm)
Maxillary and mandibular anteroposterior measurements | 6 months
  They will be measured on CBCT by linear and angular measurements(mm and angles)
Vertical skeletal measurents | 6 months
  They will be measured on CBCT by linear and angular measurements(mm and angles)